CLINICAL TRIAL: NCT04068376
Title: Double-task Exercise Programs to Strengthen Cognitive and Vascular Health in Older Adults at Risk of Cognitive Decline: a Randomized Clinical Trial
Brief Title: Double-task Exercise in Older Adults at Risk of Cognitive Decline (MeMo-Health-Cog-3 Program)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: School of Health and Sport Sciences, Chukyo University, Japan. (Unknown); Facultad de Estudios Superiores Aragón UNAM (Unknown); university of chukyo (Unknown); Faculty of Higher Studies UNAM (Unknown)
Responsible Party: Principal Investigator, Dr. Rosalinda Sanchez Arenas, Investigator in Epidemiology, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-785-095; 2023-3-146 (Other Grant/Funding Number: INSTITUTO MEXICANO DEL SEGURO SOCIAL)
Record Dates: First submitted 2019-08-07; First posted 2019-08-28 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Decline; Vascular Health
Keywords: cognitive decline; double task; older adults
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Movement

STUDY DESIGN:
Intervention Model Description: A double-blind randomized clinical trial entitled "Mind and Movement: Towards the Cognitive Health of Older Adults" will be conducted. The study will include two intervention groups and one control group: (1) a double-task exercise program with a squared mat led by a coach (a health professional) for 24 weeks (T1-GR); (2) the same exercise program led by a coach (a health professional) for 12 weeks and then led by caregivers of older adults for another 12 weeks (T2-GR); and (3) a control group of an aerobic-balance-stretching exercise program led by a coach for 24 weeks (C-GR).
Who Masked: Participant, Investigator
Masking Description: To ensure that the groups are balanced regarding varying levels of education, study participants were not stratified and randomly allocated in blocks of four to one of the intervention groups or the control group. An independent researcher who will not participate in the study will use the Random Allocation Software to generate the allocation sequence.31 Each stratum will have its own seed. This researcher will generate uniform random integers to create the allocation order within each block. She will hold the randomization file on her computer and will give out the allocations of individual participants one at a time to the three groups. The allocations will be concealed from participants and the study staff involved in enrollment and baseline evaluation.
  The recruitment and application of the intervention for groups 1 and 2 in stages, first in Care Unit 1 and then in Care Unit 10.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (C-GR) (Active Comparator): Control group of an aerobic-balance-stretching exercise program led by a coach for 24 weeks (C-GR).
  Interventions: Other: "Mind and Movement for Cognitive Health in the Older Adult"; Other: Double-task exercise by older adults and their caregivers
- T1-GR training sessions by health professional (Experimental): The T1-GR will consist of 60-minute training sessions delivered three days a week during a 24-week period. Each session will be guided by a health professional with a nursing background previously certified to coach SSE trainings by the Institute of Square-Stepping Exercise in Mie, Japan (Chief Tomohiro Okura and Overseas Director Professor Ryosuke Shigematsu).
  Interventions: Other: Control excercise
- T2-GR older adults and their caregivers (Experimental): In the case of T2-GR, older adults and their caregivers will participate in the same SSE program led by a coach for 12 weeks; older adults will then be asked to continue SSE at home under the supervision and with the active participation of their caregivers for another 12 weeks. They will be asked to practice SSE for 60 minutes, three times a week, and to reach a ≥65% heart rate increase. In the field of sports, the people who perform the above-mentioned activities are called "pacers," and they supervise physical activity through active accompaniment of older adults.
  Interventions: Other: Control excercise

INTERVENTIONS:
Other: Control excercise — Each session will be for 60 minutes, 3 days a week, for 24 weeks. The make-up of each session is 1) 5 minutes of warm-up; 2) 30 minutes of moderate-to-strong intensity aerobic exercise, 3) 5 minutes of aerobic cool-down, 4) 20 minutes of balance-stretching exercise; and 5) 5 minutes of cool-down stretching (this times does not count as activity).
  Other Names: Aerobic-balance-stretching exercise program
  Arms: T1-GR training sessions by health professional; T2-GR older adults and their caregivers
Other: "Mind and Movement for Cognitive Health in the Older Adult" — The T1-GR will consist of 60-minute training sessions delivered three days a week during a 24-week period. Each session will be guided by a health profesional certified to coach SSE. The make-up of each session is: 1) 5 minutes of warm-up; 2) 30 minutes of moderate-to-strong intensity aerobic exercise, 3) 5 minutes of aerobic cool-down, 4) 20 minutes of double-task exercise (mat); and 5) 5 minutes of cool-down stretching (this times does not count as activity).
  Other Names: Double-task exercise by a health professional
  Arms: Control group (C-GR)
Other: Double-task exercise by older adults and their caregivers — In the case of T2-GR, older adults and their caregivers will participate in the same SSE program led by a coach for 12 weeks; older adults will then be asked to continue SSE at home under the supervision and with the active participation of their caregivers for another 12 weeks. They will be asked to practice SSE for 60 minutes, three times a week, and to reach a ≥65% heart rate increase. In the field of sports, the people who perform the above-mentioned activities are called "pacers," and they supervise physical activity through active accompaniment of older adults.
  Arms: Control group (C-GR)

SUMMARY:
Cerebral small vessel disease is a frequent cause of cognitive disability among older adults (OAs) in Mexico that imposes a significant burden on the health system and OAs' families. We have called the program Mind and Movement for Cognitive Health (MeMo-Salud-Cog-3). Programs to prevent or delay OAs' cognitive decline are scarce. Methods and analysis: A double-blind, randomized clinical trial will be conducted. The study will aim to evaluate two 24-week double-task (aerobic and cognitive) square-stepping exercise programs for OAs at risk of cognitive decline-one program with and another without caregiver participation-and to compare these with an aerobic-balance-stretching exercise program (control group). 255 OAs (85 per group) affiliated with the Mexican Institute of Social Security (IMSS) between 60 and 65 years of age with self-reported cognitive concerns will participate. They will be stratified by education level and randomly allocated to the groups. The intervention will last 24 weeks, and the effect of each program will be evaluated 12, 24, and 52 weeks after the intervention. Participants' demographic and clinical characteristics will be collected at baseline. The outcomes will include: (i) general cognitive function; (ii) specific cognitive functions; (iii) dual-task gait; (iv) blood pressure; (v) carotid intima-media thickness; (vi) carotid arterial compliance; (vii) OAs' health-related quality of life; and (viii) caregiver burden. We will estimate differences in outcomes between each intervention group and the control group at baseline and follow-up evaluations. We will assess differences-in-differences (D-in-D) treatment effects using a D-in-D estimator. If we identify statistically significant differences in participants' baseline characteristics between the groups, we will adjust the D-in-D estimators by these covariates using generalized linear regression models. Ethics and dissemination: The study was approved by the IMSS Ethics and Research Committee (registration number 2018-785-095). All participants will sign a consent form prior to their participation. The study results will be disseminated to IMSS authorities, healthcare providers and the research community.

DETAILED DESCRIPTION:
1. Aim: to evaluate two 24-week double-task (aerobic and cognitive) square-stepping exercise programs for older adults (OAs) at risk of cognitive decline - one program with and another without caregiver participation - and to compare these with an aerobic-balance-stretching exercise program (control group). 255 OAs (85 per group) affiliated with the Mexican Institute of Social Security (IMSS) between 60 and 75 years of age with self-reported cognitive concerns will participate. They will be stratified by education level and randomly allocated to the groups.
2. Study design: A double-blind randomized clinical trial entitled "Mind and Movement: Towards the Cognitive Health of Older Adults" will be conducted. The study will include two intervention groups and one control group: (1) a double-task exercise program with a squared mat led by a coach (a health professional) for 24 weeks (T1-GR); (2) the same exercise program led by a coach (a health professional) for 12 weeks and then led by caregivers of older adults for another 12 weeks (T2-GR); and (3) a control group of an aerobic-balance-stretching exercise program led by a coach for 24 weeks (C-GR).
3. Study hypothesis:

   The investigators hypothesize that T1 and T2 double-task exercise trainings will show more significant improvements in older adults than the control aerobic training with regards to (i) general cognitive function; (ii) specific cognitive functions (executive function, processing speed, verbal learning and memory, and verbal fluency); (iii) usual walking and dual-task gait; (iv) blood pressure; (v) carotid intima-media thickness; (vi) carotid arterial compliance; (vii) older adults' health-related quality of life; and (viii) caregiver burden.
4. Sample Size: It was calculated using the formula suggested by Zong (2009)32 for continuous outcome variable and non-inferiority design (2 [Z 1-α+Z 1-β/ δ] * S2). The investigators considered α <0.05, a power of 80%, and the assumptions to δ0 (a clinically acceptable margin) and S2(polled standard deviations of both comparison groups): General cognitive function=0.20(0.05), Mental flexibility (EF) part A=0.13(0.03) and B=0.37(0.37), Processing speed=0.06(0.02), Verbal learning=0.63(0.32) and memory=0.16(0.08), Verbal fluency words by category= 0.54 (0.14) and by letter=0.66 (0.17), Walking speed (cm/s)=0.23(0.06), Walking length(cm)=0.86(0.22), Systolic blood pressure(mmHg)=0.27(0.06); Diastolic blood pressure(mmHg)=0.79(0.40), Carotid intima-media thickness(mm)=0.20(0.05).Subjective burden on informal caregivers=0.53, Patient health-related quality of life (SF-36) Mental score=4.0(1.0) and Physical score=4.0(2.0). The maximum required sample size, assuming a possible 20% drop-out rate, is 85 participants per group.
5. Intervention implementation:

   The study will be conducted at IMSS Epidemiology and Health Services Research Unit facilities in Mexico City.

   The T1-GR will consist of 60-minute training sessions delivered three days a week during a 24-week period. Each session will be guided by a health professional with a nursing background previously certified to coach SSE trainings by the Institute of Square-Stepping Exercise in Mie, Japan (Chief Tomohiro Okura and Overseas Director Professor Ryosuke Shigematsu).

   In the case of T2-GR, older adults and their caregivers will participate in the same SSE program led by a coach for 12 weeks; older adults will then be asked to continue SSE at home under the supervision and with the active participation of their caregivers for another 12 weeks. They will be asked to practice SSE for 60 minutes, three times a week, and to reach a ≥65% heart rate increase. In the field of sports, the people who perform the above-mentioned activities are called "pacers," and they supervise physical activity through active accompaniment of older adults.
6. Compliance and adverse events monitoring A monitoring system will be developed to perform long-distance monitoring of compliance with physical activity. It will include three components: i) the system that will collect the information from a chipset connected to the SSE mats (e.g., time of exercise, velocity); ii) the system that will transmit and store the data on the study computer; iii) the system for supervision and follow-up, which will allow connecting with participants through different electronic devices, such as mobile phones and e-mails.

   The monitoring system will be an important strategy to avoid missing data, drop-out rates and low program adherence.

   In addition, the investigators will monitor study adverse events through direct observations of the study participants during the exercise sessions, monitoring system, and 12-, 24-, and 54-week evaluations.

   The investigators will register number, type (e.g., dizziness, pain, fatigue, muscle strains, falls, or injuries), and severity of adverse events during the exercise sessions and outside the hours of the exercise sessions but during the intervention period. The severity of events will be categorized as follows: mild (do not affect activities of daily living); moderate (have moderate effect on activities of daily living); and severe (requires hospitalization, or results in persistent or significant disability or results in some life-threatening, or other medically important condition). RSA and ABD will review all adverse events on a weekly basis. They will report all moderate and severe adverse events to the IMSS Ethics Committee and stop the study if the adverse events data demonstrate any hazard of the intervention.
7. Motivation strategies The monitoring system will be an important strategy to avoid drop-outs and low program adherence. It will be complemented by motivation phone calls to those participants who fail to attend the group sessions or to perform home-based SES activities.

   Moreover, the study will include 10-15 minute group discussions to explore health-related topics, such as the benefits of healthy lifestyles (e.g., physical activity, nutrition) to maintaining cardiovascular and brain health or to exchange experiences on past events. The discussions will precede exercise training sessions.
8. Evaluations The investigators will conduct four evaluations during the study: the baseline evaluation and 12-week, 24-week, and 52-week evaluations. The study outcome variables will be measured at each evaluation, while the covariates will be collected only at the beginning of the study. The investigators will also measure the participants' adherence to the programs, defined as 80% or higher compliance with the assigned exercise training regimen. Finally, the investigators will document the reasons for dropouts and poor adherence. Previously trained health professionals with a medical specialty in geriatrics will perform these evaluations.

   The study covariates will cover Participant demographic and clinical characteristics: age (years from birth); biological sex (male or female); formal educational attainment (years); current employment status (retired, employed, volunteer, unpaid worker, unemployed); marital status (married, widowed, divorced, single, other); and current living situation (living alone, living with a spouse, living with or without children); self-reported comorbidities relevant to this study (e.g., vascular risk factors, orthopedic conditions, etc.); and self-reported baseline physical activity defined as i) ideal (≥150 minutes per week of moderate-intensity activity or ≥75 minutes per week of vigorous-intensity activity, or an equivalent combination); ii) moderate/intermediate (≤149 minutes per week of moderate-intensity activity or ≤74 minutes per week of vigorous or intense activity, or an equivalent combination); and iii) poor (without any moderate or intense physical activity). The apolipoprotein E (APOE) ε4 allele is a genetic risk factor for Alzheimer's.

   Caregivers will be asked the following: age, biological sex, formal educational attainment, current employment status, marital status, relation to the patient, and self-reported baseline physical activity, as previously defined; availability of social support networks; and presence of animal companions at home. Social support will be measured using the Household and Family Support Networks subsection (part 5) of the World Health Organization Study on Global AGEing and Adult Health.
9. Data Management and confidentiality Data entry will be conducted by trained staff. Data quality will be assessed before statistical analysis (eg, range checks for data values).

   Only members of the study team will have access to the study information and all information that will be collected from participants will be kept private to ensure confidentiality. The consent forms with participant signatures will be stored in a locked location only accessible by the principal investigator (PI). All electronic data will be stored on the PI laptop and a back-up hard drive which will be password protected. Any handwritten information such as field notes or other related research materials will be stored and secured in a locked cabinet when not in use. Data will be erased and destroyed after 5 years, as per IMSS Ethics and Research Committee guidelines. Only deidentified data will be used for reporting, publication, and dissemination of findings.
10. Statistical Analysis First, the investigators will perform a descriptive analysis of the older adults' and caregivers' characteristics at each evaluation and evaluate the distribution of quantitative variables using the Kilmogorov-Smirnov normality test. Variables that have normal distribution will be analyzed using means and standard deviations, variables with non-normal distribution will be presented using medians and 25th and 75th percentiles, and categorical variables will be analyzed by using frequencies and percentages. Second, for each evaluation the investigators will compare study variables between T1-GR and C-GR and between T2-GR and C-GR. The comparison between these groups will be performed using Student's t-test (for normally distributed continuous variables), Mann Whitney-U test (for continuous variables that are not normally distributed), or Chi-square test (for categorical variables), as appropriate. The difference between baseline and post-intervention evaluations for each group will be measured using the Student's paired t-test or Mann-Whitney U test when the distribution is non-normal. The effect of the intervention on the outcome variables will be assessed by estimating the differences-in-differences (D-in-D) treatment effects using a D-in-D estimator.46 If the investigators identify statistically significant differences in participants' baseline characteristics and adherence to the exercise regimens among the studied groups, the model will adjust the results of the D-in-D treatment effects by these covariates using a generalized linear regression model (GLM), where Yi= ß0+ ß1Xi+ß2X+ ß3X +ßjCov +ei; in this regression equation, ß1 represents the mean difference within each group, β2 the mean change after the intervention, β3 the difference in mean change between the two groups (e.g., T1-GR and C-GR), ßjCov the covariates that were different between the study groups, and ei= the standard error. This model considers the correlation among repeated observations of the same subject and allows a more precise estimate to be obtained. The investigators will conduct a model for each outcome variables. P-values < 0.05 will be interpreted as statistically significant. The analyses will be performed using the software Stata 14.0 (Stata Corp, College Station, TX, USA).

ELIGIBILITY:
Inclusion criteria.

1. With 60-75 years of age.
2. They have self-reported cognitive concerns (ie, have answered "yes" to the question: "Do you feel like your memory or thinking skills have gotten worse recently?").
3. They demonstrate functional independence in activities of daily living and instrumental activities of daily living.
4. They have one or more vascular risk factors (eg, type 2 diabetes or hypertension).
5. They have symptoms or signs of underlying cognitive dysfunction without a diagnosis of dementia (ie, confirmed by a review of their health records and a Mini Mental State Exam [MMSE] score> 24).
6. They have an informal caregiver who accepts to participate.

Exclusion criteria.

1. With depression (score> 15 according to the Center for Epidemiological Studies Depression Scale - Revised [CESD-R]).
2. With clinically significant neurological or psychiatric disorders (eg, Parkinson's, schizophrenia).
3. With a recent severe cardiovascular event (eg, myocardial infarction, stroke).
4. With a major orthopedic condition (eg, severe osteoarthritis).
5. With blood pressure that is unsafe for exercise (ie,> 180/100 mmHg or <100/60 mmHg).
6. With a severe visual or auditory impairment.
7. With an unwillingness to adhere to the intervention schedules.

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
General Cognitive funtion | 0 weeks
  i) Subjective memory complaints were evaluated through five questions: "Do you have difficulty remembering things?" "Do you feel as though you have forgotten conversations?" "Have you asked the same question several times?" "Have you recently forgotten to turn off the stove?" "Do you think you have memory problems?" Each affirmative response was scored one point, while a negative response received zero points. Therefore, the minimum possible score was zero, and the maximum was five points. ii) The Mini-Mental State Examination (MMSE) uses a 0 to 30-point scale to identify mild cognitive impairment. iii) The Montreal Cognitive Assessment (MoCA), also on a 0 to 30-point scale. iv) The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) assesses cognitive function through 11 items related to memory, language, praxis, and orientation, providing a comprehens cognitive assessment, with total scores ranging from 0 to 69.
General Cognitive funtion | 24 weeks
  i) Subjective memory complaints were evaluated through five questions: "Do you have difficulty remembering things?" "Do you feel as though you have forgotten conversations?" "Have you asked the same question several times?" "Have you recently forgotten to turn off the stove?" "Do you think you have memory problems?" Each affirmative response was scored one point, while a negative response received zero points. Therefore, the minimum possible score was zero, and the maximum was five points. ii) The Mini-Mental State Examination (MMSE) uses a 0 to 30-point scale to identify mild cognitive impairment. iii) The Montreal Cognitive Assessment (MoCA), also on a 0 to 30-point scale. iv) The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) assesses cognitive function through 11 items related to memory, language, praxis, and orientation, providing a comprehensive cognitive assessment, with total scores ranging from 0 to 69.
General Cognitive funtion | 52 weeks
  i) Subjective memory complaints were evaluated through five questions: "Do you have difficulty remembering things?" "Do you feel as though you have forgotten conversations?" "Have you asked the same question several times?" "Have you recently forgotten to turn off the stove?" "Do you think you have memory problems?" Each affirmative response was scored one point, while a negative response received zero points. Therefore, the minimum possible score was zero, and the maximum was five points. ii) The Mini-Mental State Examination (MMSE) uses a 0 to 30-point scale to identify mild cognitive impairment. iii) The Montreal Cognitive Assessment (MoCA), also on a 0 to 30-point scale. iv) The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) assesses cognitive function through 11 items related to memory, language, praxis, and orientation, providing a comprehens cognitive assessment, with total scores ranging from 0 to 69.
Specific domains of cognitive function | 0 weeks
  Measured through composite scores: Executive function/mental flexibility will be measured with the Trail Making Tests, Part A and Part B. The results for both TMT-A and TMT-B are reported as the number of seconds required to complete a task. Processing speed (using the Digit Symbol Substitution Test) will be measured as the total correct number-symbol matches achieved in 90 seconds. Verbal learning and memory will be assessed through Rey's Auditory Verbal Learning Test (RAVLT) that consists of documenting the number of words remembered from a list of 15 words presented in two separate moments; this test allows evaluation of the RAVLT-Immediate and RAVLT-Percent Forgetting. Verbal fluency (semantic, animal naming, and phonemic) will be measured by using the Controlled Oral Word Association Test and assessed through the total number of words identified by category and letter. The frontal assessment battery (FAB)
Specific domains of cognitive function | 24 weeks
  Measured through composite scores: Executive function/mental flexibility will be measured with the Trail Making Tests, Part A and Part B. The results for both TMT-A and TMT-B are reported as the number of seconds required to complete a task. Processing speed (using the Digit Symbol Substitution Test) will be measured as the total correct number-symbol matches achieved in 90 seconds. Verbal learning and memory will be assessed through Rey's Auditory Verbal Learning Test (RAVLT) that consists of documenting the number of words remembered from a list of 15 words presented in two separate moments; this test allows evaluation of the RAVLT-Immediate and RAVLT-Percent Forgetting. Verbal fluency (semantic, animal naming, and phonemic) will be measured by using the Controlled Oral Word Association Test and assessed through the total number of words identified by category and letter.
Specific domains of cognitive function | 52 weeks
  Measured through composite scores: Executive function/mental flexibility will be measured with the Trail Making Tests, Part A and Part B. The results for both TMT-A and TMT-B are reported as the number of seconds required to complete a task. Processing speed (using the Digit Symbol Substitution Test) will be measured as the total correct number-symbol matches achieved in 90 seconds. Verbal learning and memory will be assessed through Rey's Auditory Verbal Learning Test (RAVLT) that consists of documenting the number of words remembered from a list of 15 words presented in two separate moments; this test allows evaluation of the RAVLT-Immediate and RAVLT-Percent Forgetting. Verbal fluency (semantic, animal naming, and phonemic) will be measured by using the Controlled Oral Word Association Test and assessed through the total number of words identified by category and letter.
Cognitive reserve | 0 weeks
  Capacity that enables an individual to cope with and/or recover from the impact of a neural injury or a psychotic episode.
Cognitive reserve | 24 weeks
  Capacity that enables an individual to cope with and/or recover from the impact of a neural injury or a psychotic episode.
Cognitive reserve | 52 weeks
  Capacity that enables an individual to cope with and/or recover from the impact of a neural injury or a psychotic episode.

SECONDARY OUTCOMES:
Usual walking and dual-task gait | 0 weeks
  Usual walking and dual-task gait will be evaluated through motion capture during the six-minute walk test (6MWT), which requires participants to walk back and forth across a 30-metre area at a comfortable pace for six minutes. The fixed distance utilized by 6MWT allows determination of gait speed (i.e., v=d/t); however, this test will also be coupled with infrared stride analysis, which will allow for a more precise evaluation of gait speed, stride length, and stride variability under usual and dual-task conditions. These procedures will provide a number of valid and reliable gait outcomes through the synchronization of mobility data via eight infrared cameras, six force plates, and electromyography.
Usual walking and dual-task gait | 24 weeks
  Usual walking and dual-task gait will be evaluated through motion capture during the six-minute walk test (6MWT), which requires participants to walk back and forth across a 30-metre area at a comfortable pace for six minutes. The fixed distance utilized by 6MWT allows determination of gait speed (i.e., v=d/t); however, this test will also be coupled with infrared stride analysis, which will allow for a more precise evaluation of gait speed, stride length, and stride variability under usual and dual-task conditions. These procedures will provide a number of valid and reliable gait outcomes through the synchronization of mobility data via eight infrared cameras, six force plates, and electromyography.
Usual walking and dual-task gait | 52 weeks
  Usual walking and dual-task gait will be evaluated through motion capture during the six-minute walk test (6MWT), which requires participants to walk back and forth across a 30-metre area at a comfortable pace for six minutes. The fixed distance utilized by 6MWT allows determination of gait speed (i.e., v=d/t); however, this test will also be coupled with infrared stride analysis, which will allow for a more precise evaluation of gait speed, stride length, and stride variability under usual and dual-task conditions. These procedures will provide a number of valid and reliable gait outcomes through the synchronization of mobility data via eight infrared cameras, six force plates, and electromyography.
Carotid intima-media thickness (cIMT) | 0 weeks
  Carotid intima-media thickness (cIMT) is the thickness of the two innermost layers of the arterial wall, intima and median in cm and will be measured through an ultrasound of the right common carotid artery. Specifically, a longitudinal B-mode image (Philips HDI 5000 ultrasound, 7-12 MHz linear array transducer) of the cephalic portion of the right common carotid artery will be obtained by a trained ultrasound technician. The composite IMT was calculated as the means of near and far wall IMT of all carotid segments, millimeters.
Carotid intima-media thickness (cIMT) | 24 weeks
  Carotid intima-media thickness (cIMT) is the thickness of the two innermost layers of the arterial wall, intima and median in cm and will be measured through an ultrasound of the right common carotid artery. Specifically, a longitudinal B-mode image (Philips HDI 5000 ultrasound, 7-12 MHz linear array transducer) of the cephalic portion of the right common carotid artery will be obtained by a trained ultrasound technician. The composite IMT was calculated as the means of near and far wall IMT of all carotid segments, millimeters.
Carotid intima-media thickness (cIMT) | 52 weeks
  Carotid intima-media thickness (cIMT) is the thickness of the two innermost layers of the arterial wall, intima and median in cm and will be measured through an ultrasound of the right common carotid artery. Specifically, a longitudinal B-mode image (Philips HDI 5000 ultrasound, 7-12 MHz linear array transducer) of the cephalic portion of the right common carotid artery will be obtained by a trained ultrasound technician. The composite IMT was calculated as the means of near and far wall IMT of all carotid segments, millimeters.
Quality of life as measured by SF-12 | 0 weeks
  Older adults' health-related quality of life (QoL) will be measured by the short form (SF-12) of the Medical Outcomes Survey questionnaire, comprised of 12 items. Physical and mental scores will be calculated using an algorithm to convert each item response into standardized values according to specific predetermined weights. Summary scores for each component range from 0-100 and are interpreted as low QoL (close to 0) and high QoL (approaching 100).
Quality of life as measured by SF-12 | 24 weeks
  Older adults' health-related quality of life (QoL) will be measured by the short form (SF-12) of the Medical Outcomes Survey questionnaire, comprised of 12 items. Physical and mental scores will be calculated using an algorithm to convert each item response into standardized values according to specific predetermined weights. Summary scores for each component range from 0-100 and are interpreted as low QoL (close to 0) and high QoL (approaching 100).
Quality of life as measured by SF-12 | 52 weeks
  Older adults' health-related quality of life (QoL) will be measured by the short form (SF-12) of the Medical Outcomes Survey questionnaire, comprised of 12 items. Physical and mental scores will be calculated using an algorithm to convert each item response into standardized values according to specific predetermined weights. Summary scores for each component range from 0-100 and are interpreted as low QoL (close to 0) and high QoL (approaching 100).
Subjective Caregiver Burden | 0 weeks
  Subjective burden on informal caregivers will be measured using the short form of the Burden Scale for Family Caregivers (BSFC-s)-a 10-item instrument. Each item is measured on a four-point scale with the values "strongly disagree" (0), "disagree" (1), "agree" (2), and "strongly agree" (3). A high degree of agreement indicates higher perception of burden by the caregiver.
Subjective Caregiver Burden | 24 weeks
  Subjective burden on informal caregivers will be measured using the short form of the Burden Scale for Family Caregivers (BSFC-s)-a 10-item instrument. Each item is measured on a four-point scale with the values "strongly disagree" (0), "disagree" (1), "agree" (2), and "strongly agree" (3). A high degree of agreement indicates higher perception of burden by the caregiver.
Subjective Caregiver Burden | 52 weeks
  Subjective burden on informal caregivers will be measured using the short form of the Burden Scale for Family Caregivers (BSFC-s)-a 10-item instrument. Each item is measured on a four-point scale with the values "strongly disagree" (0), "disagree" (1), "agree" (2), and "strongly agree" (3). A high degree of agreement indicates higher perception of burden by the caregiver.
Cardiovascular biomarkers and endothelial function: MCP-1, ICAM VCAM and Selectin | 0 weeks
  This is the ability of circulating vascular cell adhesion molecule-1 (VCAM-1), endothelial-leukocyte adhesion molecule-1 (E-selectin), and intercellular adhesion molecule-1 (ICAM-1) to serve as molecular markers of atherosclerosis and predictors of incident cardiovascular disease.
Cardiovascular biomarkers and endothelial function: MCP-1, ICAM VCAM and Selectin | 24 weeks
  This is the ability of circulating vascular cell adhesion molecule-1 (VCAM-1), endothelial-leukocyte adhesion molecule-1 (E-selectin), and intercellular adhesion molecule-1 (ICAM-1) to serve as molecular markers of atherosclerosis and predictors of incident cardiovascular disease.
Cardiovascular biomarkers and endothelial function: MCP-1, ICAM VCAM and Selectin | 52 weeks
  This is the ability of circulating vascular cell adhesion molecule-1 (VCAM-1), endothelial-leukocyte adhesion molecule-1 (E-selectin), and intercellular adhesion molecule-1 (ICAM-1) to serve as molecular markers of atherosclerosis and predictors of incident cardiovascular disease.
Holter | 0 weeks
  Holter will be measured as part of the monitoring system. Participants will be provided with an appropriately sized ambulatory Holter monitoring device.
  This is a cardiology study that records the heart's electrical activity for 24 hours or more, allowing the doctor to analyze the heart rhythm during the patient's daily activities.
Holter | 24 weeks
  Holter will be measured as part of the monitoring system. Participants will be provided with an appropriately sized ambulatory Holter monitoring device.
  This is a cardiology study that records the heart's electrical activity for 24 hours or more, allowing the doctor to analyze the heart rhythm during the patient's daily activities.
Holter | 52 weeks
  Holter will be measured as part of the monitoring system. Participants will be provided with an appropriately sized ambulatory Holter monitoring device.
  This is a cardiology study that records the heart's electrical activity for 24 hours or more, allowing the doctor to analyze the heart rhythm during the patient's daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalinda Sánchez Arenas, PhD, Study Director — Instituto Mexicano del Seguro Socil
Locations (1):
- Rosalinda Sánchez Arenas, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mimenza-Alvarado A, Aguilar-Navarro SG, Yeverino-Castro S, Mendoza-Franco C, Avila-Funes JA, Roman GC. Neuroimaging Characteristics of Small-Vessel Disease in Older Adults with Normal Cognition, Mild Cognitive Impairment, and Alzheimer Disease. Dement Geriatr Cogn Dis Extra. 2018 May 16;8(2):199-206. doi: 10.1159/000488705. eCollection 2018 May-Aug. PMID 29928288
- [Result] Shigematsu R, Okura T. A novel exercise for improving lower-extremity functional fitness in the elderly. Aging Clin Exp Res. 2006 Jun;18(3):242-8. doi: 10.1007/BF03324655. PMID 16804371
- [Result] Verghese J, LeValley A, Hall CB, Katz MJ, Ambrose AF, Lipton RB. Epidemiology of gait disorders in community-residing older adults. J Am Geriatr Soc. 2006 Feb;54(2):255-61. doi: 10.1111/j.1532-5415.2005.00580.x. PMID 16460376
- [Result] Inzitari M, Metti A, Rosano C, Udina C, Perez LM, Carrizo G, Verghese J, Newman AB, Studenski S, Rosso AL. Qualitative neurological gait abnormalities, cardiovascular risk factors and functional status in older community-dwellers without neurological diseases: The Healthy Brain Project. Exp Gerontol. 2019 Sep;124:110652. doi: 10.1016/j.exger.2019.110652. Epub 2019 Jul 6. PMID 31288087
- [Result] Trujillo AJ, Mroz TA, Piras C, Angeles G, Tran N. Caregiving and elderly health in Mexico. Int J Health Serv. 2012;42(4):667-94. doi: 10.2190/HS.42.4.f. PMID 23367799
- [Result] Orgeta V, Miranda-Castillo C. Does physical activity reduce burden in carers of people with dementia? A literature review. Int J Geriatr Psychiatry. 2014 Aug;29(8):771-83. doi: 10.1002/gps.4060. PMID 25191688
- [Result] Gregory MA, Boa Sorte Silva NC, Gill DP, McGowan CL, Liu-Ambrose T, Shoemaker JK, Hachinski V, Holmes J, Petrella RJ. Combined Dual-Task Gait Training and Aerobic Exercise to Improve Cognition, Mobility, and Vascular Health in Community-Dwelling Older Adults at Risk for Future Cognitive Decline1. J Alzheimers Dis. 2017;57(3):747-763. doi: 10.3233/JAD-161240. PMID 28304305
- [Result] Boa Sorte Silva NC, Gregory MA, Gill DP, McGowan CL, Petrella RJ. The Impact of Blood Pressure Dipping Status on Cognition, Mobility, and Cardiovascular Health in Older Adults Following an Exercise Program. Gerontol Geriatr Med. 2018 Apr 23;4:2333721418770333. doi: 10.1177/2333721418770333. eCollection 2018 Jan-Dec. PMID 29761133
- [Result] Gregory MA, Gill DP, Zou G, Liu-Ambrose T, Shigematsu R, Fitzgerald C, Hachinski V, Shoemaker K, Petrella RJ. Group-based exercise combined with dual-task training improves gait but not vascular health in active older adults without dementia. Arch Gerontol Geriatr. 2016 Mar-Apr;63:18-27. doi: 10.1016/j.archger.2015.11.008. Epub 2015 Dec 2. PMID 26791167
- [Result] Kramer AF, Colcombe S. Fitness Effects on the Cognitive Function of Older Adults: A Meta-Analytic Study-Revisited. Perspect Psychol Sci. 2018 Mar;13(2):213-217. doi: 10.1177/1745691617707316. PMID 29592650
- [Result] Baker LD, Frank LL, Foster-Schubert K, Green PS, Wilkinson CW, McTiernan A, Plymate SR, Fishel MA, Watson GS, Cholerton BA, Duncan GE, Mehta PD, Craft S. Effects of aerobic exercise on mild cognitive impairment: a controlled trial. Arch Neurol. 2010 Jan;67(1):71-9. doi: 10.1001/archneurol.2009.307. PMID 20065132
- [Result] Lautenschlager NT, Cox KL, Flicker L, Foster JK, van Bockxmeer FM, Xiao J, Greenop KR, Almeida OP. Effect of physical activity on cognitive function in older adults at risk for Alzheimer disease: a randomized trial. JAMA. 2008 Sep 3;300(9):1027-37. doi: 10.1001/jama.300.9.1027. PMID 18768414
- [Result] Middleton L, Kirkland S, Rockwood K. Prevention of CIND by physical activity: different impact on VCI-ND compared with MCI. J Neurol Sci. 2008 Jun 15;269(1-2):80-4. doi: 10.1016/j.jns.2007.04.054. Epub 2008 Feb 20. PMID 18243244
- [Result] Kelly ME, Loughrey D, Lawlor BA, Robertson IH, Walsh C, Brennan S. The impact of cognitive training and mental stimulation on cognitive and everyday functioning of healthy older adults: a systematic review and meta-analysis. Ageing Res Rev. 2014 May;15:28-43. doi: 10.1016/j.arr.2014.02.004. Epub 2014 Mar 4. PMID 24607830
- [Result] Willis SL, Tennstedt SL, Marsiske M, Ball K, Elias J, Koepke KM, Morris JN, Rebok GW, Unverzagt FW, Stoddard AM, Wright E; ACTIVE Study Group. Long-term effects of cognitive training on everyday functional outcomes in older adults. JAMA. 2006 Dec 20;296(23):2805-14. doi: 10.1001/jama.296.23.2805. PMID 17179457
- [Result] Klusmann V, Evers A, Schwarzer R, Schlattmann P, Reischies FM, Heuser I, Dimeo FC. Complex mental and physical activity in older women and cognitive performance: a 6-month randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2010 Jun;65(6):680-8. doi: 10.1093/gerona/glq053. Epub 2010 Apr 23. PMID 20418350
- [Result] Holtzer R, Verghese J, Xue X, Lipton RB. Cognitive processes related to gait velocity: results from the Einstein Aging Study. Neuropsychology. 2006 Mar;20(2):215-23. doi: 10.1037/0894-4105.20.2.215. PMID 16594782
- [Result] Springer S, Giladi N, Peretz C, Yogev G, Simon ES, Hausdorff JM. Dual-tasking effects on gait variability: the role of aging, falls, and executive function. Mov Disord. 2006 Jul;21(7):950-7. doi: 10.1002/mds.20848. PMID 16541455
- [Result] Verghese J, Robbins M, Holtzer R, Zimmerman M, Wang C, Xue X, Lipton RB. Gait dysfunction in mild cognitive impairment syndromes. J Am Geriatr Soc. 2008 Jul;56(7):1244-51. doi: 10.1111/j.1532-5415.2008.01758.x. Epub 2008 May 14. PMID 18482293
- [Result] Montero-Odasso M, Muir SW, Speechley M. Dual-task complexity affects gait in people with mild cognitive impairment: the interplay between gait variability, dual tasking, and risk of falls. Arch Phys Med Rehabil. 2012 Feb;93(2):293-9. doi: 10.1016/j.apmr.2011.08.026. PMID 22289240
- [Result] Cheng ST. Cognitive Reserve and the Prevention of Dementia: the Role of Physical and Cognitive Activities. Curr Psychiatry Rep. 2016 Sep;18(9):85. doi: 10.1007/s11920-016-0721-2. PMID 27481112
- [Result] Shigematsu R, Okura T, Nakagaichi M, Tanaka K, Sakai T, Kitazumi S, Rantanen T. Square-stepping exercise and fall risk factors in older adults: a single-blind, randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2008 Jan;63(1):76-82. doi: 10.1093/gerona/63.1.76. PMID 18245764
- [Result] Gates N, Fiatarone Singh MA, Sachdev PS, Valenzuela M. The effect of exercise training on cognitive function in older adults with mild cognitive impairment: a meta-analysis of randomized controlled trials. Am J Geriatr Psychiatry. 2013 Nov;21(11):1086-97. doi: 10.1016/j.jagp.2013.02.018. Epub 2013 Jul 3. PMID 23831175
- [Result] Cabanero-Martinez MJ, Cabrero-Garcia J, Richart-Martinez M, Munoz-Mendoza CL. [Structured review of activities of daily living measures in older people]. Rev Esp Geriatr Gerontol. 2008 Sep-Oct;43(5):271-83. doi: 10.1016/s0211-139x(08)73569-8. Spanish. PMID 18842201
- [Result] Kohout FJ, Berkman LF, Evans DA, Cornoni-Huntley J. Two shorter forms of the CES-D (Center for Epidemiological Studies Depression) depression symptoms index. J Aging Health. 1993 May;5(2):179-93. doi: 10.1177/089826439300500202. PMID 10125443
- [Result] Zhong B. How to calculate sample size in randomized controlled trial? J Thorac Dis. 2009 Dec;1(1):51-4. PMID 22263004
- [Result] Gill DP, Gregory MA, Zou G, Liu-Ambrose T, Shigematsu R, Hachinski V, Fitzgerald C, Petrella RJ. The Healthy Mind, Healthy Mobility Trial: A Novel Exercise Program for Older Adults. Med Sci Sports Exerc. 2016 Feb;48(2):297-306. doi: 10.1249/MSS.0000000000000758. PMID 26285025
- [Result] Farran CJ, Paun O, Cothran F, Etkin CD, Rajan KB, Eisenstein A, Navaie M. Impact of an Individualized Physical Activity Intervention on Improving Mental Health Outcomes in Family Caregivers of Persons with Dementia: A Randomized Controlled Trial. AIMS Med Sci. 2016;3(1):15-31. doi: 10.3934/medsci.2016.1.15. Epub 2015 Dec 17. PMID 29147683
- [Result] Mollinedo Cardalda I, Lopez A, Cancela Carral JM. The effects of different types of physical exercise on physical and cognitive function in frail institutionalized older adults with mild to moderate cognitive impairment. A randomized controlled trial. Arch Gerontol Geriatr. 2019 Jul-Aug;83:223-230. doi: 10.1016/j.archger.2019.05.003. Epub 2019 May 8. PMID 31100545
- [Result] Aguilar-Navarro SG, Mimenza-Alvarado AJ, Palacios-Garcia AA, Samudio-Cruz A, Gutierrez-Gutierrez LA, Avila-Funes JA. Validity and Reliability of the Spanish Version of the Montreal Cognitive Assessment (MoCA) for the Detection of Cognitive Impairment in Mexico. Rev Colomb Psiquiatr (Engl Ed). 2018 Oct-Dec;47(4):237-243. doi: 10.1016/j.rcp.2017.05.003. Epub 2017 Jul 29. English, Spanish. PMID 30286846
- [Result] Gaudino EA, Geisler MW, Squires NK. Construct validity in the Trail Making Test: what makes Part B harder? J Clin Exp Neuropsychol. 1995 Aug;17(4):529-35. doi: 10.1080/01688639508405143. PMID 7593473
- [Result] Rosano C, Perera S, Inzitari M, Newman AB, Longstreth WT, Studenski S. Digit Symbol Substitution test and future clinical and subclinical disorders of cognition, mobility and mood in older adults. Age Ageing. 2016 Sep;45(5):688-95. doi: 10.1093/ageing/afw116. Epub 2016 Jul 4. PMID 27496932
- [Result] Moradi E, Hallikainen I, Hanninen T, Tohka J; Alzheimer's Disease Neuroimaging Initiative. Rey's Auditory Verbal Learning Test scores can be predicted from whole brain MRI in Alzheimer's disease. Neuroimage Clin. 2016 Dec 18;13:415-427. doi: 10.1016/j.nicl.2016.12.011. eCollection 2017. PMID 28116234
- [Result] Malek-Ahmadi M, Small BJ, Raj A. The diagnostic value of controlled oral word association test-FAS and category fluency in single-domain amnestic mild cognitive impairment. Dement Geriatr Cogn Disord. 2011;32(4):235-40. doi: 10.1159/000334525. Epub 2011 Dec 8. PMID 22156335
- [Result] Graessel E, Berth H, Lichte T, Grau H. Subjective caregiver burden: validity of the 10-item short version of the Burden Scale for Family Caregivers BSFC-s. BMC Geriatr. 2014 Feb 20;14:23. doi: 10.1186/1471-2318-14-23. PMID 24555474
- [Result] Dhamoon MS, Dong C, Elkind MS, Sacco RL. Ideal cardiovascular health predicts functional status independently of vascular events: the Northern Manhattan Study. J Am Heart Assoc. 2015 Feb 12;4(2):e001322. doi: 10.1161/JAHA.114.001322. PMID 25677566
- [Result] Parra-Rodriguez L, Gonzalez-Meljem JM, Gomez-Dantes H, Gutierrez-Robledo LM, Lopez-Ortega M, Garcia-Pena C, Medina-Campos RH. The Burden of Disease in Mexican Older Adults: Premature Mortality Challenging a Limited-Resource Health System. J Aging Health. 2020 Aug-Sep;32(7-8):543-553. doi: 10.1177/0898264319836514. Epub 2019 Mar 27. PMID 30913945
- [Result] Perez-Cuevas R, Doubova SV, Bazaldua-Merino LA, Reyes-Morales H, Martinez D, Karam R, Gamez C, Munoz-Hernandez O. A social health services model to promote active ageing in Mexico: design and evaluation of a pilot programme. Ageing Soc. 2015 Aug;35(7):1457-1480. doi: 10.1017/S0144686X14000361. Epub 2014 May 23. PMID 26190874
- [Result] Dao E, Hsiung GR, Liu-Ambrose T. The role of exercise in mitigating subcortical ischemic vascular cognitive impairment. J Neurochem. 2018 Mar;144(5):582-594. doi: 10.1111/jnc.14153. Epub 2017 Sep 27. PMID 28833160
- [Result] Lambert SD, Bowe SJ, Livingston PM, Heckel L, Cook S, Kowal P, Orellana L. Impact of informal caregiving on older adults' physical and mental health in low-income and middle-income countries: a cross-sectional, secondary analysis based on the WHO's Study on global AGEing and adult health (SAGE). BMJ Open. 2017 Nov 15;7(11):e017236. doi: 10.1136/bmjopen-2017-017236. PMID 29146639
- [Result] Jacob L, Oh H, Shin JI, Haro JM, Vancampfort D, Stubbs B, Jackson SE, Smith L, Koyanagi A. Informal Caregiving, Chronic Physical Conditions, and Physical Multimorbidity in 48 Low- and Middle-Income Countries. J Gerontol A Biol Sci Med Sci. 2020 Jul 13;75(8):1572-1578. doi: 10.1093/gerona/glaa017. PMID 31943005
- [Derived] Sanchez-Arenas R, Doubova SV, Bernabe-Garcia M, Gregory MA, Mejia-Alonso LA, Orihuela-Rodriguez O, Paredes-Manjarrez C, Colin-Martinez T, Mujica-Morales I, Grijalva-Otero I, Basurto-Acevedo L, Manuel-Apolinar L, Cuadros-Moreno J, Bernal-Diaz A, Shigematsu R. Double-task exercise programmes to strengthen cognitive and vascular health in older adults at risk of cognitive decline: protocol for a randomised clinical trial. BMJ Open. 2020 Dec 30;10(12):e039723. doi: 10.1136/bmjopen-2020-039723. PMID 33380479
- See also: Instituto Mexicano del Seguro Social. Informe al Ejecutivo Federal y al Congreso de la Unión Sobre la situación financiera y los riesgos del Instituto Mexicano del Seguro Social 2017-2018. — http://www.imss.gob.mx/sites/all/statics/pdf/informes/20172018/21-InformeCompleto.pdf
- See also: Prueba de caminata de 6 minutos: recomendaciones y procedimientos. — https://www.medigraphic.com/pdfs/neumo/nt-2015/nt152h.pdf
- See also: Consejo Nacional de Población. La situación demográfica de México 2017 (text in Spanish). — https://www.gob.mx/conapo/documentos/la-situacion-demografica-de-mexico-2017?idiom=es
- See also: Envejecimiento y dependencia. Realidades y previsión para los próximos años. — https://www.anmm.org.mx/publicaciones/CAnivANM150/L11-Envejecimiento-y-dependencia.pdf